CLINICAL TRIAL: NCT02894567
Title: Evaluation of Directional Recording and Stimulation Using the spiderSTN During the Implantation of DBS Leads
Brief Title: Evaluation of Directional Recording and Stimulation Using spiderSTN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was structured in 2 phases, and was stopped after the first phase. The collected data will be used to improve the device and prepare future studies.
Sponsor: Aleva Neurotherapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KEK 272-15; CIV-16-02-014704 (Other: EUDAMED)
Record Dates: First submitted 2016-08-24; First posted 2016-09-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Parkinson's Disease; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- spiderSTN (Experimental): It is an Intraoperative test during a deep brain stimulation surgery. The spiderSTN lead is implanted in a selected track in the brain, and is tested for stimulation and recording.
  Interventions: Device: Intraoperative test during a deep brain stimulation surgery

INTERVENTIONS:
Device: Intraoperative test during a deep brain stimulation surgery — The spiderSTN lead is inserted in a selected track in the brain, and is connected to external neuro-recorder/stimulator . Once the intraoperative test phase is completed, the test devices are removed and the DBS surgery resumes.

SUMMARY:
The purpose of this study is to provide proof-of-concept that directional stimulation and directional recording, in an intraoperative setting, is perceivable in a subject. The tests will be performed using a dedicated intraoperative lead connected to an external neuro-recorder/stimulator, during a deep brain stimulation implantation surgery.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) technique involves implanting electrodes using a stereotactic method and connecting them to a pulse generator to deliver a current in localized areas in the brain.

The optimum location for DBS electrodes is determined by pre-operative brain imaging, often combined with an intraoperative microelectrode recording/stimulating (MER) sequence. Current MER practice involves inserting micro-recording/stimulating electrodes into guide tubes in the brain and lowering them towards the target, performing recordings at selected steps. The recordings differ based on the types of neuronal structures they are passing through.Based on the recordings, some promising locations are further discriminated by stimulation using macro-electrodes, and the target for final lead placement is chosen.

The spiderSTN lead (Aleva Neurotherapeutics SA, Switzerland) is capable of recording and stimulating from both its inner and outer surface, allowing the user to steer the direction of stimulation during the target location phase. This will allow the neurosurgeon greater flexibility in investigating the balance between therapeutic benefits and stimulation-induced side effects at a given location.

This feasibility study is designed to explore the effect of directional stimulation and the ability to differentiate between stimulation induced side effects at a given location, during the DBS surgery. It will be proposed to patients who suffer from Parkinson disease (PD) or essential tremor (ET) and for whom DBS is indicated according to standard criteria at the hospital. It will be restricted to a limited number of patients (10), sufficient to assess the recording and stimulating capacity of the spiderSTN device. The patient undergoes the normal DBS surgery until the position for the final lead has been chosen. Then the spiderSTN test phase takes place. Once test phase is completed, the conventional DBS surgery resumes.

ELIGIBILITY:
Inclusion Criteria:

Patient foreseen to undergo DBS for Parkinson's disease or Essential Tremor according to routine criteria of the center.

For Parkinson Disease:

* Person is between 18 and 75 years of age
* Established diagnosis of idiopathic Parkinson's disease with progression of symptoms for a minimum of 2 years.
* Person has a history of at least 30% improvement on the UPDRS therapy in L-dopa (levodopa), except in the case of tremor dominant patient
* Weak control of symptoms by dopaminergic therapy (off phenomenon, fluctuations on / off, dyskinesia on)

For Essential Tremor:

* Person is between 18 and 80 years of age
* Established diagnosis of Essential Tremor for a minimum of 2 years
* Functional disability due to tremor was not adequately controlled by medication for at least 3 months prior to implant.

Person has given his/her written consent

Exclusion Criteria:

* Person suffering from an active major psychiatric disorder
* Mattis Dementia Rating Scale score <130 or otherwise not capable of discernment
* Presence of major co-morbidity or medical condition that may affect participation to the study
* Presence of an electrical or electromagnetic implant (e.g., cochlear implant, pacemaker)
* Person with a previous surgery for the treatment of Parkinson's disease or Essential Tremor
* Person with a previous brain ablation procedure
* Person who suffers from epilepsy
* Person who is pregnant: a pregnancy test will be performed in patients of childbearing age
* Person with coagulopathies
* Abuse of drugs or alcohol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Measurement of the delivered electrical current at which a sustained side effect occurs, and compare the results from specific angular directions | up to one hour during surgery
  This will be performed by independently stimulating electrodes which are oriented in different directions on the same spiderSTN lead, and assessing the patient's response.

SECONDARY OUTCOMES:
Measurement of the electrical current created by the neuronal activity coming from specific directions, and compare the results. | up to one hour during surgery
  To assess the recording capabilities of the spiderSTN lead by correlating the results obtained from the neurologist's visual, real-time interpretation of the recorded neuronal activity, to a post-processing analysis of the actual signal recorded.
Electrical functionality of the study device during the test phase | 1 day
  The electrical integrity of the device will be measured before and after the test phase, to confirm that it was functional throughout the test phase.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Pollo, Professor, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided